CLINICAL TRIAL: NCT04562194
Title: NEVA ONE One-Pass Reperfusion With the NeVa Stent-Retriever EMEA Registry
Brief Title: NeVa ONE Registry Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-003/D
Record Dates: First submitted 2020-09-04; First posted 2020-09-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Thrombus; stroke
MeSH Terms: conditions — Ischemic Stroke; Thrombosis; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Other): NeVa Stent Retriever
  Interventions: Device: NeVa Stent Retriever

INTERVENTIONS:
Device: NeVa Stent Retriever — mechanical neurothrombectomy

SUMMARY:
A prospective, open label study designed to assess the safety, performance and efficacy of thrombus removal in subjects presenting with acute ischemic stroke with the NeVa stent retrievers.

DETAILED DESCRIPTION:
This is a prospective, open label, multi-center registry designed to assess the safety, performance and efficacy of the NeVa stent retriever in the treatment of large vessel occlusion strokes. Up to 600 subjects will be enrolled at up 30 sites.

ELIGIBILITY:
Inclusion Criteria:

Only subjects already treated with the NeVa thrombectomy devices can be considered for enrollment.

1. Age ≥18
2. NIHSS score ≥ 6
3. Pre-stroke mRS score ≤ 1
4. Intracranial arterial occlusion of the distal intracranial carotid artery or middle cerebral artery (M1/M2), anterior cerebral artery (ACA), posterior cerebral artery (PCA), basilar artery, or vertebral artery demonstrated with DSA.
5. Thrombectomy procedure can be initiated within 24 hours from symptom onset (defined as time last known well [TLKW])
6. Imaging Inclusion Criteria:

   The patient should have confirmed LVO and salvageable penumbra. Any automated software for determine the volume of viable tissue is acceptable. patient selection should follow the following guidelines:
   * ASPECTS 6-10 if treatment started 0-6 hours from TLKW
   * ASPECTS 8-10 if treatment started 6-24 hours from TLKW
   * Ischemic core ≤ 50 cc
7. Subject or legal representative is able and willing to give informed consent within 72 hours after the intervention (may use independent physician consent in this timeframe and gain subject or legal representative consent later than 72 hours).

Exclusion Criteria:

1. Pre-existing medical neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept).
2. Cardiopulmonary resuscitation, significant cardiac arrhythmia, evidence of ongoing myocardial infarction, concern for pre- treatment pulmonary aspiration.
3. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories
4. Cerebral vasculitis
5. History of severe allergy to contrast medium.
6. Known allergy to NeVa materials (nitinol, stainless steel)
7. Suspicion of aortic dissection, septic embolus, or bacterial endocarditis
8. Systemic infection
9. Significant mass effect with midline shift
10. Evidence of intracranial tumor (except small meningioma)
11. Inability to deploy NeVA device for at least one pass for any other reason
12. Life expectancy less than 6 months
13. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
First Pass Success Rate | post-procedure day 0
  The primary study endpoint is the first pass success rate with the NeVa device defined as eTICI score ≥ 2B & eTICI ≥2C

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Espanol de Mendoza, Mendoza, Argentina
- Niguarda Hospital, Milan, Italy
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates